CLINICAL TRIAL: NCT01853371
Title: The Efficacy of Wet Cupping on Blood Pressure Among Hypertension Patients in Jeddah, 2013, A Pilot Study
Brief Title: Efficacy of Wet Cupping on Blood Pressure Among Hypertension Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Collaborators: Joint Program of Family and Community Medicine, Jeddah, Saudi Arabia (Other); King Fahd Medical Research Centre (Other)
Responsible Party: Principal Investigator, Nouran Aleyeidi, Community Medicine PHD Candidate, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2013-05-07; First posted 2013-05-15 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wet cupping and conventional treatment (Experimental): Wet cupping: Will be administered through 3 sessions, with 4 weeks interval between each session and the other.
  Conventional treatment: Is the usual anti-HTN treatment taken by the patients at the King Abdulaziz university hospital outpatient department.
  Interventions: Procedure: Wet cupping; Other: Conventional treatment
- Conventional treatment (Active Comparator): Conventional treatment: Is the usual anti-HTN treatment taken by the patients at the King Abdulaziz university hospital outpatient department.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Procedure: Wet cupping — Wet cupping is the process of using a vacuum at different points on the body in order to gather the blood in that area. Then apply few superficial incisions (small, light scratches using a razor) on those areas, followed by repeating the vacuum on the same areas in order to remove 'harmful' blood which lies just beneath the surface of the skin. In this study, the wet cupping procedure was not done on certain days of the lunar month.
  Other Names: Hijama
  Arms: Wet cupping and conventional treatment
Other: Conventional treatment — According to Saudi Hypertension management guidelines, hypertension patients may require life style modification alone , especially for newly diagnosed cases, or my require life style modification and drug treatment. This will be decided by the treating team in the hospital.
  Other Names: Anti-hypertension management

SUMMARY:
This research proposal is submitted to fulfill the requirement of the PHD degree of Community Medicine Saudi Board at the Joint Program of Family and Community Medicine in Jeddah, Saudi Arabia.

Background: Cupping is an ancient treatment remedy that has been used for many centuries in many parts of the world. In the Middle East, Wet cupping "Hijama" is still a popular treatment because of its religious background. Despite of that, it still has little scientific evidence that proves its efficacy. Many hijama healers claim that they have observed dramatic improvement in Blood pressure control of hypertension patients. Not many studies support that. This study should help to prove or disprove this hypothesis.

Objectives:

* To determine the efficacy of wet cupping on blood pressure among high blood pressure patients.
* To assess the incidence of wet cupping side effects in the intervention group.

Methods: The study design is a randomised controlled trial. There will be an intervention group of high blood pressure patients who will perform hijama in addition to their usual management, and a control group of high blood pressure patients who will receive their usual anti-hypertension management only. There will be 4 weeks follow up period. After that, data entry, analysis and interpretation will take place.

Hypothesis: Wet cupping has an effect on blood pressure in adult hypertension patients

ELIGIBILITY:
Inclusion Criteria:

* High BP at the time of the study (SBP 140 mmHg or more and/or DBP 90mmHg or more). For patients with DM, high BP is defined as SBP 130 mmHg or more and/or DBP 85mmHg or more.
* Age between 19 and 65 years old.
* Males and females

Exclusion Criteria:

* Grade III Hypertension (SBP 180 mmHg or more and/or DBP 110 BP or more).
* Patients with very high added risk,according to the Saudi Hypertension management guidelines. By excluding the patient who have associated clinical conditions which are: cerebrovascular disease, heart disease, renal disease, peripheral vascular disease and advanced retinopathy.
* Patients with secondary hypertension.
* Pregnant women.
* If the patient performed dry cupping, wet cupping or acupuncture during the past 6 months.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nouran A Aleyeidi, Resident Community Medicine, Principal Investigator — Ministry of Health; Khaled Aseri, Consultant Community Medicine, Study Director — National Guard Health Affairs, King Abdulaziz Medical City
Locations (1):
- King Abdulaziz University Hospital, Jeddah, Western Region, Saudi Arabia

RESULTS

PARTICIPANT FLOW:
Groups:
- Wet Cupping and Conventional Treatment: Wet cupping: Will be administered through 3 sessions, with 4 weeks interval between each session and the other. The wet cupping procedure was not done on certain days of the lunar month.
  Conventional treatment: Is the usual anti-HTN treatment taken by the patients at the King Abdulaziz university hospital outpatient department.
  Wet cupping: Wet cupping is the process of using a vacuum at different points on the body in order to gather the blood in that area. Then apply few superficial incisions (small, light scratches using a razor) on those areas, followed by repeating the vacuum on the same areas in order to remove 'harmful' blood which lies just beneath the surface of the skin.
  Conventional treatment: According to Saudi Hypertension management guidelines, hypertension patients may require life style modification alone , especially for newly diagnosed cases, or my require life style modification and drug treatment. This will be decided by the treating team in the hospital.
Period: Overall Study
Arm/Group | Wet Cupping and Conventional Treatment | Conventional Treatment
Started | 10 | 10
Completed | 10 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Wet Cupping and Conventional Treatment: Wet cupping: Will be administered through 3 sessions, with 4 weeks interval between each session and the other.
  Conventional treatment: Is the usual anti-HTN treatment taken by the patients at the King Abdulaziz university hospital outpatient department.
  Wet cupping: Wet cupping is the process of using a vacuum at different points on the body in order to gather the blood in that area. Then apply few superficial incisions (small, light scratches using a razor) on those areas, followed by repeating the vacuum on the same areas in order to remove 'harmful' blood which lies just beneath the surface of the skin. In this study, the wet cupping procedure was not done on certain days of the lunar month.
  Conventional treatment: According to Saudi Hypertension management guidelines, hypertension patients may require life style modification alone , especially for newly diagnosed cases, or my require life style modification and drug treatment.
- Total: Total of all reporting groups
Arm/Group | Wet Cupping and Conventional Treatment | Conventional Treatment | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.20 (7.22) | 49.43 (9.50) | 51.06 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 4 | 3 | 7
Basline Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 160.1 (13.5) | 149.4 (11.1) | 155.3 (13.3)
Baseline Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 90.6 (10.3) | 93.5 (10.6) | 91.9 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure After 4 Weeks
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Wet Cupping and Conventional Treatment | Conventional Treatment
Number analyzed (Participants) | 10 | 8
mmHg | 158.3 (15.9) | 138.9 (12.8)

2. Secondary Outcome: Incidence of Wet Cupping Side Effects in Intervention Group
Description: * Immediate side effects of wet cupping will be assessed through a checklist on the after each cupping session.
  * Delayed side effects of wet cupping will be assessed through another checklist after 1 month of the final hijama session.
Time Frame: 1 month
Reporting Status: Not Posted

3. Primary Outcome: Diastolic Blood Pressure After 4 Weeks
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Wet Cupping and Conventional Treatment | Conventional Treatment
Number analyzed (Participants) | 10 | 8
mmHg | 91 (9.3) | 88 (11.0)

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Wet Cupping and Conventional Treatment | Conventional Treatment
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8
Other Adverse Events (participants affected / at risk) | 4/10 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wet Cupping and Conventional Treatment (N=10) | Conventional Treatment (N=8)
Dizziness (General disorders) | 3 (4) | 0 (0) — appeared immediately after wet cupping session and lasted maximum for 1 day
Headache (General disorders) | 2 (2) | 0 (0)
Bullae formation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — dissappeared after 1 week
Itching at the site of wet cupping (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No